CLINICAL TRIAL: NCT02576626
Title: The Effectiveness of Single Dose Ultibro Breezhaler (Indacaterol/Glycopyrronium) by Sd-DPI Versus Ipratropium/Salbutamol by Nebulizer in Improving FEV1 and Dyspnea During Stable State of COPD
Brief Title: Single Dose Ultibro Breezhaler by Sd-DPI Versus Ipratropium/Salbutamol by Nebulizer in COPD
Acronym: ULT01
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wouter H. van Geffen (Other)
Collaborators: Novartis (Industry); University Medical Center Groningen (Other)
Responsible Party: Sponsor-Investigator, Wouter H. van Geffen, Arts onderzoeker, Groningen Research Institute for Asthma and COPD
Organization: Groningen Research Institute for Asthma and COPD (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL5250604215
Record Dates: First submitted 2015-08-04; First posted 2015-10-15 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: COPD
Keywords: Nebulizer; DPI; COPD; indacaterol; ipratropium; glycopyrronium; salbutamol; Breezhaler; Nebuliser; Hyperinflation; Dyspnea; SABA; short-acting muscarinic antagonists (SAMA); long-acting beta2-agonist (LABA); LAMA; FEV1
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — indacaterol; Ipratropium; Albuterol, Ipratropium Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Other): Participants start with Ultibro (indacaterol/glycopyrronium 110/50) + placebo nebulization , then after a new washout period of 7 days they will receive ipratropium/salbutamol nebulization and placebo Breezhaler Interventions: indacaterol/glycopyrronium 110/50 Breezhaler® ,Placebo by Breezhaler®, ipratropium/salbutamol 0,5 mg, 2,5 mg by nebulisation, Placebo by nebulisation
  Interventions: Drug: indacaterol/glycopyrronium 110/50 Breezhaler®; Device: Placebo by Breezhaler®; Drug: ipratropium/salbutamol 0,5 mg, 2,5 mg by nebulisation; Device: Placebo by nebulisation
- B (Other): Participants start with ipratropium/salbutamol nebulization and placebo Breezhaler , then after a new washout period of 7 days they will receive Ultibro(indacaterol/glycopyrronium 110/50) + placebo nebulization.
  Interventions: indacaterol/glycopyrronium 110/50 Breezhaler® ,Placebo by Breezhaler®, ipratropium/salbutamol 0,5 mg, 2,5 mg by nebulisation, Placebo by nebulisation
  Interventions: Drug: indacaterol/glycopyrronium 110/50 Breezhaler®; Device: Placebo by Breezhaler®; Drug: ipratropium/salbutamol 0,5 mg, 2,5 mg by nebulisation; Device: Placebo by nebulisation

INTERVENTIONS:
Drug: indacaterol/glycopyrronium 110/50 Breezhaler®
  Other Names: Ultibro
Device: Placebo by Breezhaler®
Drug: ipratropium/salbutamol 0,5 mg, 2,5 mg by nebulisation
  Other Names: Combivent
Device: Placebo by nebulisation

SUMMARY:
Rationale:

Inhaled bronchodilators, beta-2-agonist or anticholinergic or combinations, can be delivered by several types of devices: dry powder (DPI), pressurized metered dose inhalers (pMDI), and wet nebulizers. Wet nebulization is available for short-acting bronchodilators only, is cumbersome, and, importantly, has never been scientifically been proven to be more efficacious than delivery by the other two methods. Yet many patients are happy with wet nebulization and in many clinics this administration method prevails. The investigators believe that combined long-acting bronchodilators, are more efficacious than combined short acting bronchodilators per nebulizers.

Objective:

To test the hypothesis that: The combination of the two long-acting bronchodilators indacaterol and glycopyrronium by dry powder inhalation confers a superior improvement compared to nebulisation with ipratropium/salbutamol, when administered as single dose in patients with stable state chronic obstructive pulmonary disease (COPD).

Study design: Investigator initiated, randomised, active controlled, cross-over double-blind (and therefore double-dummy), study comparing the effects of single dose indacaterol/glycopyrronium 110/50 Breezhaler® versus single dose ipratropium/salbutamol nebulisation in patients with COPD in stable state Study population: Patients visiting the outpatient clinics or from general practitioner (GP) practices with COPD GOLD stage A-D, and (FEV1) post-bronchodilator FEV1/ forced vital capacity (FVC) < 70%; post-br FEV1 < 80%pred. Intervention The investigators will compare the effects of single dose indacaterol/glycopyrronium 110/50 Breezhaler® versus single dose ipratropium/salbutamol nebulisation in patients with COPD in stable state

Main study parameters/endpoints:

Area under the curve (AUC) from 0 to 6 hours of FEV1 with indacaterol and glycopyrronium, compared to nebulisation with ipratropium/salbutamol

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

This study has no specific benefits for the participating patients. The study also has no major risks. Minor risks for participants after a single dosis can be throat irritation, cough, headache and dizziness, sinus tachycardia. The combination of treatments with β2-agonist bronchodilators and anticholinergic bronchodilators have been used in daily practice for many years in many countries and they are often prescribed both in COPD. Both indacaterol/glycopyrronium and ipratropium/salbutamol are approved for COPD treatment in the Netherlands

ELIGIBILITY:
Inclusion Criteria:

1. COPD, post-bronchodilator FEV1/FVC < 70%; post-br FEV1 < 80%pred
2. Active mastery of Dutch
3. Written informed consent
4. At least 40 years old
5. Participants must be able to understand and complete protocol requirements, Instructions, and questionnaires provided in Dutch

Exclusion Criteria:

1. Non invasive ventilation
2. Saturation by pulse oxymetry <88%
3. Documented history of asthma
4. Instable cardiac disease within 6 months.
5. Known long corrected QT interval (QTC) syndrome
6. Known estimated Glomerular Filtration Rate (EGFR) ( <30 ml/min *1,73m2
7. Exacerbations of COPD or change of medication for COPD in the last 6 weeks prior to inclusion
8. Allergic reaction or intolerance for a substance used in one of the products or atropine or atropine derived substances
9. Pregnant or lactating females.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-12; Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of FEV1 | from 0 to 6 hours
  Area under the curve (AUC) from 0 to 6 hours of FEV1 with indacaterol and glycopyrronium, compared to nebulisation with ipratropium/salbutamol.

SECONDARY OUTCOMES:
Change in Borg dyspnea score at 30 min | 30 min up to 360 minutes
  1. Change in Borg dyspnea score at 30 min: change in Borg score at other time points
Proportion of patients reaching the minimal clinically important difference (MCID) at all time points | all time points (15, 30, 60, 120 240 and 360 min)
  proportion of patients reaching the MCID at all time points (15, 30, 60, 120 240 and 360 min) (1)
Changes in level of hyperinflation (by IC measurement) | all time points (15, 30, 60, 120 240 and 360 min)
Time to FEV1 increase of 100 ml | all time points (15, 30, 60, 120 240 and 360 min)
Peak effect of FEV1 | from 0 to 6 hours
  Maximum FEV1 per group, calculated using the best FEV1 per participant
Time to peak of FEV1 | all time points (15, 30, 60, 120 240 and 360 min)
FEV1 | at all time points (15, 30, 60, 120 240 and 360 min)
Proportion of participants reaching a difference of 100 ml of inspiratory capacity (IC) | Time Frame: all time points (15, 30, 60, 120 240 and 360 min)

CONTACTS AND LOCATIONS:
Overall Officials: Huib AM Kerstjens, prof. dr., Principal Investigator — Groningen Research Institute for Asthma and COPD; Wouter H van Geffen, MD, Study Director — Frisius Medisch Centrum
Locations (1):
- UMCG, Groningen, Netherlands